CLINICAL TRIAL: NCT05913362
Title: IVUS Based Ultra-low Volume Contrast Media PCI to Reduce Contrast Induced Nephrology in Patient With Chronic Kidney disease-a Multi-center, Open Label, Randomized Trial (IVUS-CKD)
Brief Title: IVUS Guided PCI for CKD to Reduce CI-AKI
Acronym: IVUS-CKD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jilin University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Zhongnan Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other); The Sixth People's Hospital of Zhengzhou (Other); China-Japan Union Hospital, Jilin University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Mingyou Zhang, Associate prof, Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVUSCKD
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease; Chronic Kidney Diseases
Keywords: CKD; IVUS; CAD; PCI
MeSH Terms: conditions — Coronary Artery Disease; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVUS based ultra-low contrast PCI (Experimental): IVUS based ultra-low contrast PCI
  Interventions: Behavioral: IVUS based ultralow contrast PCI
- Standard of care PCI (No Intervention): Guideline directed contrast induced nephropathy provention strategy with standard of care PCI procedure.

INTERVENTIONS:
Behavioral: IVUS based ultralow contrast PCI — IVUS based ultralow contrast PCI
  Arms: IVUS based ultra-low contrast PCI

SUMMARY:
Patients with Chronic kidney disease are most vulnerable to contrast induced nephropathy after Percutaneous coronary intervention, intravascular ultrasound guidance can be used to safely guide the procedure to reduce the contrast usage, this randomized trial is design to test the hypothesis that IVUS based ultra-low contrast PCI is feasible and can reduce the contrast induced nephropathy.

DETAILED DESCRIPTION:
Prospective, open-label, randomized(1:1), multi-center trial of 320 patients allocated to one of the treatment arms(IVUS-guided ultra-low contrast PCI or angiography-guided PCI).

The study population will be composed of patients with renal dysfunction referring for PCI on one to more coronary artery. target lesion must be assessable with IVUS.

eGFR will be re-evaluated 48 hours after the procedure. and at 1 month, 3 month, 6 month, 12 month. as well as follow-up for other clinical outcomes unless contra-indicated all patients will receive intravenous hydration 12 hours before and after the procedure. saline infusion at a dose of 1ml/kg/hour. if with reduced ejection fraction or overt heart failure reduce the saline infusion to 0.5ml/kg/hour. the use of sodium bicarbonate and diuretic will be left at the discretion of the operator All procedure will be performed using non-ionic, low osmolar or iso-osmolar, iodine-based contrast media the study groups will be compared according to the intention-to-treat principle. Categorial variables will be compared by Fisher's exact test and continuous variables by students T test. Time-dependent events will be estimated by the Kaplan-Meier method and compared by hazards cox model or log-rank test.

ELIGIBILITY:
Inclusion Criteria:

- age over 18 years coronary artery disease referred for percutaneous intervention, with stent, Drug coated bloon, or bioresorbable stent, of one or more epicardial vessel.

target lesion must be assessable by IVUS at baseline and during the procedure. 60ml/min/1.73m2<=Baseline Calculated creatinine clearance >=15ml/min/1.73m2 consent can be obtained and comply with all study procedures.

Exclusion Criteria:

- Use of >50ml of iodinated agent<72 hours Planned used of iodinated contrast within 72 hours after the index procedure use of other nephrotoxic agents<7 days known allergy to contrast agents unstable or unknown renal function prior to PCI life expectancy less than 1 year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Contrast-induced acute kidney injury | within 72 hours after the index procedure (or at discharge).
  Evaluate whether IVUS-guided PCI reduces CI-AKI. CI-AKI defined as an increase in serum creatine>=0.5mg
  /dl from the baseline, within 72 hours after the index procedure(or at discharge) comparison to stand-alone angiography-guided PCI. CI-AKI will be defined as an increase in serum creatinine ≥ 0.3 mg/dl （26.52umol）from the baseline value

SECONDARY OUTCOMES:
Major adverse cardiac events and components | 1 year
  cardiovascular death, myocardial infarction and target vessel Revascularization
stent thrombosis | 1 year
  stents thrombosis will be defines as the occurrence of definite or probably stent thrombosis according to the ARC criteria
serious acute kidney dysfunction | 1 year
  >=2mg
  /dl increase of serum creatine or need for dialysis
procedure time | 1 day
  procedure time from gain access to finish the procedure
radiation exposure | 1 day
  total radiation exposure dose

CONTACTS AND LOCATIONS:
Overall Officials: Mingyou Zhang, Principal Investigator — Jilin University
Locations (2):
- China (2):
  - Jilin university, Changchun, Jilin
  - Zhongshan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCullough PA, Choi JP, Feghali GA, Schussler JM, Stoler RM, Vallabahn RC, Mehta A. Contrast-Induced Acute Kidney Injury. J Am Coll Cardiol. 2016 Sep 27;68(13):1465-1473. doi: 10.1016/j.jacc.2016.05.099. PMID 27659469
- [Background] Rudnick MR, Leonberg-Yoo AK, Litt HI, Cohen RM, Hilton S, Reese PP. The Controversy of Contrast-Induced Nephropathy With Intravenous Contrast: What Is the Risk? Am J Kidney Dis. 2020 Jan;75(1):105-113. doi: 10.1053/j.ajkd.2019.05.022. Epub 2019 Aug 28. PMID 31473019
- [Background] Mariani J Jr, Guedes C, Soares P, Zalc S, Campos CM, Lopes AC, Spadaro AG, Perin MA, Filho AE, Takimura CK, Ribeiro E, Kalil-Filho R, Edelman ER, Serruys PW, Lemos PA. Intravascular ultrasound guidance to minimize the use of iodine contrast in percutaneous coronary intervention: the MOZART (Minimizing cOntrast utiliZation With IVUS Guidance in coRonary angioplasTy) randomized controlled trial. JACC Cardiovasc Interv. 2014 Nov;7(11):1287-93. doi: 10.1016/j.jcin.2014.05.024. Epub 2014 Oct 15. PMID 25326742